CLINICAL TRIAL: NCT03997721
Title: Pathophysiology of Perioperative Fluid Management in Patients Un-dergoing High Risk Emergency Laparotomy, a Prospective Descriptive Cohort Study
Brief Title: Pathophysiology of Perioperative Fluid Management in Emergency Laparotomy
Status: Completed | Type: Observational
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Mirjana Cihoric, MD, Research fellow, Copenhagen University Hospital, Hvidovre
Other Study IDs: H-19010653
Record Dates: First submitted 2019-05-23; First posted 2019-06-25 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Intestinal Obstruction; Intestinal Perforation; Anastomotic Leak; Fluid Overload; Pathophysiology
Keywords: emergency laparotomy; ileus; perforated ulcer; intestinal perforation; perioperative fluid management; pathophysiology; fluid overload
MeSH Terms: conditions — Intestinal Obstruction; Intestinal Perforation; Anastomotic Leak; Edema; Ileus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Perforation: Patients undergoing primary emergency laparotomy/laparoscopy due to suspicion of intestinal perforation or ( small intestine, large intestine), perforated ventricular or duodenal ulcer
- Obstruction: Patients undergoing primary emergency laparotomy/laparoscopy due to suspicion of intestinal obstruction
- Anasomotic leak: Patients undergoing primary emergency laparotomy/laparoscopy due to suspicion of anastomotic leak following elective surgery.

SUMMARY:
Pathophysiology of perioperative fluid management in patients undergoing emergency laparotomy.

DETAILED DESCRIPTION:
In critically ill patients and patients undergoing major surgery, the combination of internal fluid shifts and fluid retention resulting in extravascular fluid accumulation and postoperative organ dysfunctions, complicates perioperative fluid management and influences patient outcome.

Changes in extravascular volume after surgery have been much debated, studies in major surgery suggest that extracellular volume expansion may correlate with intraoperative fluid administration, while other studies show the intravascular volume to be decreased after surgery.

Difficulty in obtaining accurate measurements of the fluid phases is recognized and despite years of research, perioperative extravascular volume changes have not been clarified in acute high-risk abdominal (AHA) surgery. It is essential to be able to identify and characterize the transition from necessary fluid resuscitation to harmful fluid volume accumulation, intra- as well as extravascular.

The present study seeks to investigate the perioperative fluid status and fluid shifts in patients undergoing AHA surgery, specifically focusing on intra- versus extra-vascular fluid status in patients with intestinal obstruction versus intestinal perforation.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (18 years or over) undergoing emergency high-risk abdominal surgery for following abdominal pathology:

   1. Perforated small intestine
   2. Perforated large intestine
   3. Perforated ulcer
   4. Intestinal obstruction
   5. Anastomotic leakage following elective surgery
2. Provided verbal and written informed consent
3. Must speak and understand the Danish language

Exclusion Criteria:

1. Appendectomies, cholecystectomies, negative diagnostic laparoscopies/laparotomies, herniotomies without bowel resections, sub-acute internal hernias after gastric bypass surgery, sub-acute surgery for inflammatory bowel diseases.
2. Primary surgery for intestinal ischemia, abdominal bleed
3. Emergency re-operations after elective surgery owing to intraabdominal bleeding, paralytic/obstructive ileus, intestinal ischemia
4. Reoperation owing to fascial separation with no other abdominal pathology identified and sub-acute colorectal cancer-surgery were excluded from the cohort. Sub-acute surgery was defined as surgery planned within 48 hours.
5. Traumas, gynecological, urogenital and other vascular pathology, pregnant patients.
6. Dementia and/or cognitive dysfunction (diagnosed).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults (18 years or over) undergoing emergency high-risk abdominal surgery on suspicion of intestinal perforation (incl. ulcer), obstruction, anastomotic leak.
Sampling Method: Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2019-05-23 (Actual); Primary Completion 2021-03-02 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
The fluid distribution, during the early perioperative period (≤ 5 days), in patients with intestinal perforation versus intestinal obstruction versus postoperative complications with peritonitis. | perioperative period
  Intra vs. extra vascular. Stroke volume assessment, Bioimpedance measurements

SECONDARY OUTCOMES:
Impact of fluid distribution/fluid overload on preload dependency. | Preoperatively, 6 hours postoperatively and on first, third and fifth postoperative day
Impact of fluid distribution/fluid overload on peripheral perfusion. | Preoperatively, 6 hours postoperatively and on first, third and fifth postoperative day
Correlation between fluid balance just prior to surgery and intraoperative need for vasopressor/inotropes administration. | Preoperatively, 6 hours postoperatively and on first, third and fifth postoperative day
Evaluate the relationship between fluid overload and mortality rate in patients undergoing emergency laparotomy. | Preoperatively, 6 hours postoperatively and on first, third and fifth postoperative day
Association between pre- to postoperative changes in volume status and perioperative fluid volume administration, in patients with intestinal perforation versus intestinal obstruction versus postoperative complications with peritonitis. | Preoperatively, 6 hours postoperatively and on first, third and fifth postoperative day

CONTACTS AND LOCATIONS:
Overall Officials: Nicolai Bang Foss, MD, DMSc, Study Chair — Department of Anesthesiology, Copenhagen University Hospital Hvidovre, Denmark
Locations (1):
- Copenhagen University Hospital Hvidovre, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cihoric M, Kehlet H, Hojlund J, Lauritsen ML, Kanstrup K, Foss NB. Perioperative changes in fluid distribution and haemodynamics in acute high-risk abdominal surgery. Crit Care. 2023 Jan 16;27(1):20. doi: 10.1186/s13054-023-04309-9. PMID 36647120